CLINICAL TRIAL: NCT04231825
Title: At-home Transcranial Alternating Current Stimulation During Multitasking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 18-26268-1
Record Dates: First submitted 2019-10-08; First posted 2020-01-18 (Actual); Results first posted 2021-10-28 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Multitasking Behavior
MeSH Terms: conditions — Multitasking Behavior | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Verum Stimulation (Experimental): This group will receive 6-Hz tACS
  Interventions: Device: Transcranial alternating current stimulation
- Frequency Control (Active Comparator): This group will receive 1-Hz tACS
  Interventions: Device: Transcranial alternating current stimulation

INTERVENTIONS:
Device: Transcranial alternating current stimulation — Transcranial alternating current stimulation across the prefrontal cortex using electrodes F3 and F4.

SUMMARY:
The goal is to replicate in-lab results from transcranial alternating current stimulation (tACS) with at-home tACS.

DETAILED DESCRIPTION:
Participants will be assessed in-lab on multitasking and sustained attention abilities. Participants will be sent home with a tACS device to be used at-home for five days while engaged in a multitasking paradigm that is different from the multitasking outcome measure used pre/post tACS. After the at-home stimulation is complete, participants return to UCSF for a final in-lab assessment of multitasking and sustained attention ability.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Grade 12 or more education
* Normal or corrected to normal vision and hearing
* Ability to complete cognitive tasks
* Ability to cooperate and comply with all study procedures
* Ability to tolerate tACS

Exclusion Criteria:

* Neurological or psychiatric disorders
* Family history of epilepsy
* History of seizures
* Prior head trauma
* Pregnant
* Implanted electronic devices (e.g., pacemaker)
* IQ < 80
* Taking psychotropic medication
* Taking anti-depressants or anti-anxiety medication
* Substance abuse
* Color blind
* Glaucoma
* Macular degeneration
* Amblyopia
* Strabismus

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2020-08-15 (Actual); Study Completion 2020-09-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Theodore Zanto, Ph.D., Principal Investigator — University of California, San Francisco
Locations (1):
- Sandler Neurosciences Center, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
The dataset includes self-reported information, behavioral and electrophysiological data. The final dataset will be stripped of identifiers prior to release for sharing, thereby anonymizing the data. We will make the anonymized data available to users only under a data-sharing agreement that provides for: (1) a commitment to using the data only for research purposes and not to attempt to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed. This will be in accordance with human subject regulations.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will be available after the results have been determined and the study researchers are unblinded. The data will be available indefinitely upon request.
Access Criteria: Contact PI.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Verum Stimulation | Frequency Control
Started | 23 | 24
Completed | 20 | 20
Not Completed | 3 | 4
Not completed — Protocol Violation | 3 | 3
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: Only data from participants who completed the full protocol were analyzed
Groups:
- Total: Total of all reporting groups
Arm/Group | Verum Stimulation | Frequency Control | Total
Number analyzed (Participants) | 23 | 24 | 47
Age, Categorical [Count of Participants; unit: Participants] — Population: Only data from participants who completed the full protocol were analyzed
  Participants
    number analyzed (Participants) | 20 | 20 | 40
    <=18 years | 1 | 1 | 2
    Between 18 and 65 years | 19 | 19 | 38
    >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Only data from participants who completed the full protocol were analyzed
  years
    number analyzed (Participants) | 20 | 20 | 40
    (all) | 25.8 (4.6) | 24.6 (4.2) | 25.2 (4.4)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Only data from participants who completed the full protocol were analyzed
  Participants
    number analyzed (Participants) | 20 | 20 | 40
    Female | 12 | 13 | 25
    Male | 8 | 7 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Only data from participants who completed the full protocol were analyzed
  Participants
    number analyzed (Participants) | 20 | 20 | 40
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 3 | 4 | 7
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 1 | 2 | 3
    White | 15 | 12 | 27
    More than one race | 1 | 2 | 3
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants] — Population: Only data from participants who completed the full protocol were analyzed
  Participants
    United States: number analyzed (Participants) | 20 | 20 | 40
    United States | 20 | 20 | 40
Single Task Performance [Mean (Standard Deviation); unit: d'] — Discrimination performance (d') was measured for each participant by comparing hit (correct responses to target signs) rates and false alarm (responses to non-targets) rates and calculated as d' = Z (hits) - Z (false alarms). Performance was collected during the single task condition. Population: Only data from participants who completed the full protocol were analyzed
  d'
    number analyzed (Participants) | 20 | 20 | 40
    (all) | 1.73 (0.63) | 2.01 (0.63) | 1.87 (0.63)
Multitask performance [Mean (Standard Deviation); unit: d'] — Discrimination performance (d') was measured for each participant by comparing hit (correct responses to target signs) rates and false alarm (responses to non-targets) rates and calculated as d' = Z (hits) - Z (false alarms). Performance was collected during the multitasking condition. Population: Only data from participants who completed the full protocol were analyzed
  d'
    number analyzed (Participants) | 20 | 20 | 40
    (all) | 1.03 (0.63) | 1.20 (0.58) | 1.12 (0.60)
Multitasking Cost Performance [Mean (Standard Deviation); unit: Percent change] — Discrimination performance (d') was measured for each participant by comparing hit (correct responses to target signs) rates and false alarm (responses to non-targets) rates and calculated as d' = Z (hits) - Z (false alarms). Ratio of d' during single task target discrimination task to multitask target discrimination, expressed as percentage. Population: Only data from participants who completed the full protocol were analyzed.
  Percent change
    number analyzed (Participants) | 20 | 20 | 40
    (all) | 45.8 (0.40) | 40.5 (0.22) | 43.2 (0.31)
Continuous Performance Task RT [Mean (Standard Deviation); unit: milliseconds] — Response times (in ms) during the continuous performance (sustained attention) task. Population: Only data from participants who completed the full protocol were analyzed
  milliseconds
    number analyzed (Participants) | 20 | 20 | 40
    (all) | 322 (43) | 322 (34) | 322 (39)
Continuous Performance Task RTV [Mean (Standard Deviation); unit: milliseconds] — Response time variability (standard deviation of response times in ms) during the continuous performance (sustained attention) task Population: Only data from participants who completed the full protocol were analyzed
  milliseconds
    number analyzed (Participants) | 20 | 20 | 40
    (all) | 76 (7) | 65 (5) | 71 (6)

OUTCOME MEASURES:

1. Primary Outcome: Multitasking Performance Cost (Neuroracer Performance Change From Baseline)
Description: Assessment of multitasking ability using change from baseline scores in d' cost (metric of discriminability). Discrimination performance (d') was measured for each participant by comparing hit (correct responses to target signs) rates and false alarm (responses to non-targets) rates and calculated as d' = Z (hits) - Z (false alarms). d' cost was then calculated as the ratio of d' during single task target discrimination task to multitask target discrimination, expressed as percentage cost.
Time Frame: Pre-tACS and post-tACS (1 week later)
Population: Only data from participants who completed the full protocol were analyzed
Measure: Mean (Standard Deviation); unit: percentage change of d'
Arm/Group | Verum Stimulation | Frequency Control
Number analyzed (Participants) | 20 | 20
percentage change of d' | 45.3 (0.31) | 37.9 (0.27)
Statistical Analysis 1: Comparison: Verum Stimulation vs Frequency Control; Test type: Superiority; p = 0.55, ANCOVA

2. Secondary Outcome: Continuous Performance Test RT Change (Test of Visual Attention / Sustained Attention)
Description: Assessment of sustained attention ability using response time (in ms) during the continuous performance test
Time Frame: Pre-tACS and post-tACS (1 week later)
Population: Only data from participants who completed the full protocol were analyzed
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Verum Stimulation | Frequency Control
Number analyzed (Participants) | 20 | 20
milliseconds | 300 (42) | 303 (31)
Statistical Analysis 1: Comparison: Verum Stimulation vs Frequency Control; Test type: Superiority; p = 0.51, ANCOVA

3. Secondary Outcome: Continuous Performance Test RTV Change (Test of Visual Attention / Sustained Attention)
Description: Assessment of sustained attention ability using response time variability (standard deviation of response times in ms) during the continuous performance test
Time Frame: Pre-tACS and post-tACS (1 week later)
Population: Only data from participants who completed the full protocol were analyzed
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Verum Stimulation | Frequency Control
Number analyzed (Participants) | 20 | 20
milliseconds | 58 (26) | 56 (21)
Statistical Analysis 1: Comparison: Verum Stimulation vs Frequency Control; Test type: Superiority; p = 0.80, ANCOVA

4. Primary Outcome: Single Task Performance Change
Description: Discrimination performance (d') was measured during single task performance for each participant by comparing hit (correct responses to target signs) rates and false alarm (responses to non-targets) rates and calculated as d' = Z (hits) - Z (false alarms). Performance data was collected during the single task condition.
Time Frame: Pre-tACS and post-tACS (1 week later)
Population: Only data from participants who completed the full protocol were analyzed
Measure: Mean (Standard Deviation); unit: d'
Arm/Group | Verum Stimulation | Frequency Control
Number analyzed (Participants) | 20 | 20
d' | 1.99 (0.94) | 2.70 (1.07)
Statistical Analysis 1: Comparison: Verum Stimulation vs Frequency Control; Test type: Superiority; p = 0.02, ANCOVA

5. Primary Outcome: Multitask Performance Change
Description: Discrimination performance (d') was measured while multitasking for each participant by comparing hit (correct responses to target signs) rates and false alarm (responses to non-targets) rates and calculated as d' = Z (hits) - Z (false alarms). Performance data was collected during the multitask condition.
Time Frame: Pre-tACS and post-tACS (1 week later)
Population: Only data from participants who completed the full protocol were analyzed
Measure: Mean (Standard Deviation); unit: d'
Arm/Group | Verum Stimulation | Frequency Control
Number analyzed (Participants) | 20 | 20
d' | 1.17 (0.76) | 1.79 (0.89)
Statistical Analysis 1: Comparison: Verum Stimulation vs Frequency Control; Test type: Superiority; p = 0.03, ANCOVA

ADVERSE EVENTS:
Time Frame: 10 months
Arm/Group | Verum Stimulation | Frequency Control
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/24
Other Adverse Events (participants affected / at risk) | 1/23 | 2/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Verum Stimulation (N=23) | Frequency Control (N=24)
Other (Not Including Serious) Adverse Event (Product Issues) | 1 (1) | 2 (2) — Device malfunction.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-08-11): https://cdn.clinicaltrials.gov/large-docs/25/NCT04231825/Prot_SAP_001.pdf
  • Informed Consent Form (2019-09-03): https://cdn.clinicaltrials.gov/large-docs/25/NCT04231825/ICF_002.pdf